CLINICAL TRIAL: NCT04397601
Title: AflibeRcept or Bevacizumab In Combination With Folfiri as Second-line Treatment of RAS Mutated metastaTIc cOlorectal Cancer patieNts
Brief Title: Aflibercept or Bevacizumab as Second-line Treatment of RAS Mutated Metastatic Colorectal Cancer
Acronym: ARBITRATION
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Cancer Institute, Naples (Other)
Responsible Party: Principal Investigator, Alessandro Ottaiano, Principal Investigator, National Cancer Institute, Naples
Other Study IDs: 04/20
Record Dates: First submitted 2020-05-13; First posted 2020-05-21 (Actual); Last update posted 2020-05-21 (Actual); Status verified 2020-05

CONDITIONS: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Bevacizumab; aflibercept

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- A: mCRC RAS mutated patients progressing to first-line chemotherapy with fluoropyrimidines, oxaliplatin and bevacizumab.
  Interventions: Drug: Folfiri/Bevacizumab
- B: mCRC RAS mutated patients progressing to first-line chemotherapy with fluoropyrimidines, oxaliplatin and bevacizumab.
  Interventions: Drug: Folfiri/Aflibercept

INTERVENTIONS:
Drug: Folfiri/Bevacizumab — Irinotecan (180 mg/m2), leucovorin (400 mg/m2), fluorouracil as an intravenous bolus of 400 mg/m2, and fluorouracil as a continuous 46-h infusion of 2400 mg/m2 in combination with bevacizumab (5 mg/kg) on day 1 of each 14-day cycle.
  Groups: A
Drug: Folfiri/Aflibercept — Irinotecan (180 mg/m2), leucovorin (400 mg/m2), fluorouracil as an intravenous bolus of 400 mg/m2, and fluorouracil as a continuous 46-h infusion of 2400 mg/m2 in combination with aflibercept (4 mg/kg) on day 1 of each 14-day cycle.
  Groups: B

SUMMARY:
Colorectal cancer is the third most frequent neoplasm after prostate and lung in man and breast and lung cancers in woman from Western Countries. The intensive study of predictive factors has strongly ameliorated the therapeutic flow-chart of metastatic colorectal cancer (mCRC) by allowing the selection of patients who benefit from specific therapies. In this context, the assessment of RAS (N- and K-) oncogene mutations is able to predict the response to anti-EGFR agents being mutated RAS mCRC patients resistant to these drugs. In this group of patients the use of anti-angiogenic drugs (bevacizumab and aflibercept) is predominant. Still to date there are no studies to guide oncologists in the selection of the best anti-angiogenic drug (bevacizumab beyond progression vs aflibercept) after failure of the first-line chemotherapy in RAS-M mCRC patients. The present is the first observational, pragmatic, prospective study aimed to report outcomes of mCRC patients treated with folfiri plus bevacizumab versus folfiri plus aflibercept in second-line treatment of mRAS mCRC. Furthermore, the serum levels of angiopoietin-1 (Ang-1), angiopoietin-2 (Ang-2), vascular endothelial growth factor-A and C (VEGF-A and C), stromal cell-derived factor-1 (SDF-1), platelet-derived growth factor beta (PDGF-β), basic fibroblast growth factor (bFGF), interleukin-8 (IL-8), chemokine (C-C motif) ligand 2 (CCL2), and chemokine (C-C motif) ligand 5 (CCL5) and Placental Growth Factor (PlGF), will be evaluated before starting second-line chemotherapy with bevacizumab or aflibercept in order to evidence any pattern related to response and/or prognosis. The hypothesis is that knowledge of eventual unbalance of these factors could help to select the best anti-angiogenic drug in second-line treatment of mRAS mCRC patients.

ELIGIBILITY:
Inclusion Criteria:

* Cytological or histological diagnosis of RAS mutated mCRC;
* progression at first-line chemotherapy with fluoropyrimidines, oxaliplatin and bevacizumab;
* stage IV;
* age <75 years;
* ECOG Performance Status 0 or 1;
* life expectancy> 3 months;
* negative pregnancy test for all potentially childbearing women.

Exclusion Criteria:

* presence of primary non-treated stenosing colorectal neoplasm;
* active or uncontrolled infections or bleedings;
* other concomitant uncontrolled diseases or blood laboratory values contraindicating the study drugs at clinician evaluation;
* presence of brain metastases;
* refusal or inability to provide informed consent;
* impossibility to guarantee follow-up.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: mCRC RAS mutated patients progressing at with first-line chemotherapy with at first-line chemotherapy based on fluoropyrimidines, oxaliplatin and bevacizumab.
Sampling Method: Probability Sample
Enrollment: 220 (Estimated)
Dates: Start 2020-05-11 (Actual); Primary Completion 2023-05-11 (Estimated); Study Completion 2024-05-11 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS). | 3 years
  OS will be measured from treatment start until death from any cause.

SECONDARY OUTCOMES:
Toxic effects. | 3 years
  Toxic effects will be assessed by CTCAE of the National Cancer Institute, version 4.0, June 14, 2010.
Responses' duration. | 3 years
  Time elapsed from date of response to progression occurrence.
Progression-free survival (PFS). | 3 years
  PFS will be determined from the date of treatment start until progression.

OTHER OUTCOMES:
Serum level of VEGF-A (Vascular Endothelial Growth Factor-A). | 3 years
  The molecule will be measured through ELISA test.
Serum level of PlGF (Placental Growth Factor). | 3 years
  The molecule will be measured through ELISA test.

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Ottaiano, MD, Principal Investigator — SSD-Innovative Therapies for Abdominal Metastases
Locations (1):
- SSD-Terapie Innovative Metastasi Addominali, Dipartimento di Oncologia Addominale, Istituto Nazionale Tumori di Napoli, IRCCS "G. Pascale"., Naples, Italy

IPD SHARING:
Plan to Share IPD: Undecided
Complete study protocol will be published.

REFERENCES:
- [Background] Ottaiano A, Capozzi M, Tafuto S, De Stefano A, De Divitiis C, Romano C, Avallone A, Nasti G. Folfiri-Aflibercept vs. Folfiri-Bevacizumab as Second Line Treatment of RAS Mutated Metastatic Colorectal Cancer in Real Practice. Front Oncol. 2019 Aug 13;9:766. doi: 10.3389/fonc.2019.00766. eCollection 2019. PMID 31456948
- [Derived] Ottaiano A, Scala S, Santorsola M, Trotta AM, D'Alterio C, Portella L, Clemente O, Nappi A, Zanaletti N, De Stefano A, Avallone A, Granata V, Notariello C, Luce A, Lombardi A, Picone C, Petrillo A, Perri F, Tatangelo F, Di Mauro A, Albino V, Izzo F, Rega D, Pace U, Di Marzo M, Chiodini P, De Feo G, Del Prete P, Botti G, Delrio P, Caraglia M, Nasti G. Aflibercept or bevacizumab in combination with FOLFIRI as second-line treatment of mRAS metastatic colorectal cancer patients: the ARBITRATION study protocol. Ther Adv Med Oncol. 2021 Mar 24;13:1758835921989223. doi: 10.1177/1758835921989223. eCollection 2021. PMID 33854566